CLINICAL TRIAL: NCT06814340
Title: "Continuous Positive Airway Pressure on Venovenous extracorporeaL Membrane Oxygenation for Acute respIratory Distress syndrOme" - CALMDOWN
Brief Title: "Continuous Positive Airway Pressure on Venovenous extracorporeaL Membrane Oxygenation for Acute respIratory Distress syndrOme"
Acronym: CALMDOWN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP230850
Record Dates: First submitted 2025-01-22; First posted 2025-02-07 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Acute Respiratory Distress Syndrome; Extracorporeal Membrane Oxygenation Complication
Keywords: ECMO; ARDS; CPAP
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group : near apneic ventilation (Experimental): Patients will received near apneic ventilation during the first 3 days of ECMO.
  Interventions: Device: ECMO + near apneic ventilation
- Standard of care : ultra-protective lung ventilation (Active Comparator): Patients will receive ultra-protective lung ventilation as it uses on usual care on ECMO.
  Interventions: Device: ECMO + ultra-protective lung ventilation

INTERVENTIONS:
Device: ECMO + near apneic ventilation — Near apneic ventilation will be use during the first 3 days of ECMO. Patients will be ventilated in BIPAP/APRV or pressure-controlled ventilation. PEEP will be set to maintain the same mean airway pressure obtained during the standardized ventilation period pre-randomization to prevent lung derecruitment (PEEP ≥15cmH2O). If BIPAP/APRV is used, an RR of 2-4/min will be set with high pressure set at 30cmH20 for 3 sec. If pressure-controlled ventilation is selected, a respiratory rate of two sigh breaths/min with 30 cmH2O plateau pressure will be applied. Each sigh breath will be of three seconds duration.
  Neuromuscular blockade and sedation could be used at the discretion of the attending physician. After 3 days on ECMO, apneic ventilation could be pursued (at the physician's discretion). If not, ultra-protective lung ventilation will be applied (i.e standard of care). Prone positioning on ECMO will be left to the physicians' discretion.
  Arms: Intervention group : near apneic ventilation
Device: ECMO + ultra-protective lung ventilation — Ultra-protective lung ventilation will be used up to the ECMO weaning. This group will receive ultra-protective lung ventilation with BIPAP/APRV or VCV mode setting a PEEP >10 cmH2O, ΔP 14-15 cmH2O, RR 15-20/min, Vt 3-4ml/kg and lowest FiO2 to maintain SpO2>92%.
  The use of prone positioning during ECMO will be left at the physician's discretion.
  Arms: Standard of care : ultra-protective lung ventilation

SUMMARY:
The CALMDOWN trial is a prospective, open-label, multicenter, comparative, controlled trial randomizing patients who received near apneic ventilation vs usual care on ECMO (ultra-protective lung ventilation).

The study goal is to investigate the benefit of early apneic ventilation in the most severe forms of acute respiratory distress syndrome (ARDS) rescued by ECMO.

Indeed, our hypothesis is that that early (near) apneic ventilation on venovenous ECMO for severe ARDS can enhance ventilator injury prevention and therefore reduce ECMO duration and mortality at Day 60.

ELIGIBILITY:
Inclusion Criteria:

1. Severe acute respiratory distress syndrome refractory to conventional therapy placed on VV-ECMO support in the 48 hours (maximum tolerance : +2h) preceding inclusion.
2. Obtain informed consent from a close relative or surrogate. According to the specifications of emergency inclusion, randomization without the close relative/surrogate consent could be performed if the patient is unable to give his/her consent and when the close relative/surrogate/family member are absent. Close relative/surrogate/family member consent will be asked as soon as possible after randomization. The patient will be asked as soon as possible to give his/her consent for the continuation of the trial when his/her condition will allow.
3. Social security registration (except AME)

Exclusion Criteria:

1. Age < 18
2. Pregnancy or breastfeeding
3. Initiation of VV-ECMO > 48 h (maximum tolerance : +2h)
4. Cardiac arrest with cumulated no flow time >10 minutes before ECMO (within 48 hours prior to inclusion)
5. Irreversible neurological pathology
6. End-stage chronic lung disease
7. Contraindications for high PEEP level: untreated pneumothorax, barotrauma
8. Irreversible ARDS with no hope for lung function recovery
9. Patient moribund on the day of randomization, SAPS II >90
10. Liver cirrhosis (Child B or C)
11. Lung transplantation
12. Burns on more than 20 % of the body surface
13. Participation in another interventional study or being in the exclusion period at the end of a previous study, expect DRESSING-ECMO trial, which evaluates the use of sterile adhesive transparent dressings impregnated with Chlorhexidine gluconate on the cumulative incidence of ECMO cannula-related infection episodes.
14. Individuals under guardianship, or permanently legally incompetent adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2029-05-06 (Estimated); Study Completion 2030-05-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the application of early apneic ventilation on four components : mortality status at D60, need for lung transplantation at D60, persisting ECMO at D60, number of days alive between randomization and day 60 without ECMO | Day 0 to Day 60
  These components will be summarized in a composite, hierarchical outcome. Each patient will be compared with every other patient in the study and assigned a score (tie: 0, win: +1, loss: -1) for each pairwise comparison based on whom fared better. If one patient survived without lung transplantation or ECMO still ongoing at day 60 and the other did not, scores of +1 and -1 will be assigned, respectively. If both patients in the pairwise comparison survived without lung transplant or ECMO still ongoing at day 60, the assigned score will depend on which patient had more days free from ECMO: the patient with more days off ECMO will receive a score of +1, while the patient with fewer days will receive a score of -1. If both patients survived and had the same number of days off ECMO, or if both patients died or had a lung transplant, they will be both assigned a score of 0 for that pairwise comparison.

SECONDARY OUTCOMES:
Mortality | From Day 1 to Day 60
  Efficacy of early apneic ventilation during VV-ECMO on mortality is defined as overall survival between inclusion and D60
Mortality | From Day 1 to Day 90
  Efficacy of early apneic ventilation during VV-ECMO on mortality is defined as overall survival between inclusion and D90
Need for lung transplant | From Day 1 to Day 60
  Efficacy of early apneic ventilation during VV-ECMO on the need for lung transplant is defined as lung transplant between inclusion and D60
Need for lung transplant | From Day 1 to Day 90
  Efficacy of early apneic ventilation during VV-ECMO on the need for a lung transplant is defined as lung transplant between inclusion and D90
Duration of ECMO support | From Day 1 to Day 60
  Defined as total duration with ECMO support between inclusion and D60
Duration of ECMO support | From Day 1 to Day 90
  Defined as total duration with ECMO support between inclusion and D90
Duration of invasive mechanical ventilation | From Day 1 to Day 60
  Defined as total duration of invasive mechanical ventilation between inclusion and D60
Duration of invasive mechanical ventilation | From Day 1 to Day 90
  Defined as total duration of invasive mechanical ventilation between inclusion and D90
Duration of Intensive Care Unit | From Day 1 to Day 60
  Defined as total duration spent in intensive care unit between inclusion and D60
Duration of Intensive Care Unit | From Day 1 to Day 90
  Defined as total duration spent in intensive care unit between inclusion and D90
Hospital length of stay | From Day 1 to Day 60
  Defined as total duration spent at the hospital between inclusion and D60
Hospital length of stay | From Day 1 to Day 90
  Defined as total duration spent at the hospital between inclusion and D90
ECMO free days | From Day 1 to Day 60
  Efficacy of early apneic ventilation during VV-ECMO on ECMO-free days is defined as the number of ECMO free-days between inclusion and D60
ECMO free days | From Day 1 to Day 90
  Efficacy of early apneic ventilation during VV-ECMO on ECMO-free days is defined as number of ECMO free-days between inclusion and D90
Invasive mechanical ventilation free days | From Day 1 to Day 60
  Efficacy of early apneic ventilation during VV-ECMO on invasive mecanical ventilation-free days between inclusion and D60
Invasive mechanical ventilation free days | From Day 1 to Day 90
  Efficacy of early apneic ventilation during VV-ECMO on invasive mecanical ventilation-free days between inclusion and D90
Renal replacement therapy-free days | From Day 1 to Day 60
  Efficacy of early apneic ventilation during VV-ECMO on renal function is defined as number of renal replacement therapy-free days between inclusion and D60
Renal replacement therapy-free days | From Day 1 to Day 90
  Efficacy of early apneic ventilation during VV-ECMO on renal function is defined as renal replacement therapy-free days between inclusion and D90
Continuous neuromuscular blockade-free days | From Day 1 to Day 60
  Efficacy of early apneic ventilation during VV-ECMO on continuous neuromuscular blockade is defined as number of continuous neuromuscular blockade-free days between inclusion and D60
Continuous neuromuscular blockade-free days | From Day 1 to Day 90
  Efficacy of early apneic ventilation during VV-ECMO on continuous neuromuscular blockade is defined as number of continuous neuromuscular blockade-free days between inclusion and D90
Intervention side effects (ventilation-associated pneumonia) | From Day 1 to Day D14
  Defined as the incidence of ventilation-associated pneumonia between inclusion and D14
Intervention side effets (need for inotropes or vasopressors) | From Day 1 to Day 14
  Defined as the incidence of need for inotropes or vasopressors within 14 days on ECMO
Intervention side effets (intravenous sedation consumption) | From Day 1 to Day 14
  Defined as the incidence of intravenous sedation consumption during the first 14 days on ECMO
Acute cor pulmonale | From Day 1 to Day 60
  Defined as the incidence of acute cor pulmonale between inclusion and D60
Acute cor pulmonale | From Day 1 to Day 90
  Defined as the incidence of acute cor pulmonale between inclusion and D90
Pneumothorax | From Day 1 to Day 60
  Defined as the incidence of pneumothorax between inclusion and D60
Pneumothorax | From Day 1 to Day 90
  Defined as the incidence of pneumothorax between inclusion and D90
Severe refractory hypoxemia on ECMO | From Day 1 to Day 60
  Defined as the incidence of refractory severe hypoxemia between inclusion and D60
Severe refractory hypoxemia on ECMO | From Day 1 to Day 90
  Defined as the incidence of refractory severe hypoxemia between inclusion and D90
Compliance of the respiratory system at D7 | From Day 1 to Day 7
  Effect of near apneic ventilation on the improvement of the compliance of the respiratory system (ml/cmH2O) at D7
Compliance of the respiratory system at D10 | From Day 1 to Day 10
  Effect of near apneic ventilation on the improvement of the compliance of the respiratory system (ml/cmH2O) at D10
Compliance of the respiratory system at D14 | From Day 1 to Day 14
  Effect of near apneic ventilation on the improvement of the compliance of the respiratory system (ml/cmH2O) at D14
Compliance of the respiratory system at D28 | From Day 1 to Day 28
  Effect of near apneic ventilation on the improvement of the compliance of the respiratory system (ml/cmH2O) at D28
Compliance of the respiratory system at D60 | From Day 1 to Day 60
  Effect of near apneic ventilation on the improvement of the compliance of the respiratory system (ml/cmH2O) at D60
Right ventricular function at D3 | From Day 1 to Day 3
  Effect of near apneic ventilation on right ventricular function evaluated by echocardiograohy (RV/LV diameter ratio) at D3 on ECMO following randomization
Right ventricular function at D7 | From Day 1 to Day 7
  Effect of near apneic ventilation on right ventricular function evaluated by echocardiograohy (RV/LV diameter ratio) at D7 on ECMO following randomization
Right ventricular function at D14 | From Day 1 to Day 14
  Effect of near apneic ventilation on right ventricular function evaluated by echocardiograohy (RV/LV diameter ratio) at D14 on ECMO following randomization
Right ventricular function at D28 | From Day 1 to Day 28
  Effect of near apneic ventilation on right ventricular function evaluated by echocardiograohy (RV/LV diameter ratio) at D28 on ECMO following randomization
Right ventricular function at D60 | From Day 1 to Day 60
  Effect of near apneic ventilation on right ventricular function evaluated by echocardiograohy (RV/LV diameter ratio) at D60 on ECMO following randomization

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Avicenne Hospital, Bobigny
  - Henri Mondor Hospital, Créteil
  - Pitié-Salpêtrière Hospital, Paris

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor.
Access Criteria: Researchers who provide a methodologically sound proposal.